CLINICAL TRIAL: NCT00714181
Title: A Phase I Study of Hydroxychloroquine in Combination With Temozolomide in Patients With Advanced Solid Tumors
Brief Title: Hydroxychloroquine and Temozolomide in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000600329; UPCC-12907
Record Dates: First submitted 2008-07-11; First posted 2008-07-14 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Hydroxychloroquine; Temozolomide; Blotting, Western; Microscopy, Electron; Chromatography, High Pressure Liquid; Immunoenzyme Techniques; Immunohistochemistry; Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: hydroxychloroquine
Drug: temozolomide
Genetic: TdT-mediated dUTP nick end labeling assay
Genetic: western blotting
Other: electron microscopy
Other: high performance liquid chromatography
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: mass spectrometry
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as hydroxychloroquine and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of hydroxychloroquine when given together with temozolomide in treating patients with metastatic or unresectable solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose (MTD) of hydroxychloroquine (HCQ) when administered in combination with temozolomide (TMZ) in patients with metastatic or unresectable solid tumors.

Secondary

* To determine the toxicity and toxicity rate of HCQ when administered at the MTD in combination with TMZ in these patients.

Tertiary

* To construct a population pharmacokinetic (PK) model using a limited sampling of whole blood to determine the drug exposure of HCQ and HCQ metabolites in these patients.
* To measure changes in autophagic vesicle accumulation by immunoblotting against the autophagy marker LC3 in protein lysates prepared from peripheral blood mononuclear cells (PBMC) collected from patients treated with HCQ and TMZ.
* To measure changes in median number of autophagic vesicles by electron microscopy in PBMC collected from patients treated with HCQ and TMZ.
* To assess tumor changes in LC3 and caspase 3 cleavage by western blotting.
* To assess tumor cell death characteristics by immunohistochemical methods (Ki67, TUNEL staining, cleaved caspase 3).
* To evaluate autophagy by electron microscopy.
* To define associations between changes in LC3 levels from baseline in PBMC with HCQ exposure.
* To measure the levels of HMGB1 in the serum of patients treated with HCQ and TMZ.

OUTLINE: This is a dose-escalation study of hydroxychloroquine (HCQ).

Patients receive oral HCQ alone once or twice daily for 14 days. Patients then receive oral HCQ once or twice daily on days 1-28 and oral temozolomide once daily on days 1-7 and 15-21. Treatment with HCQ and temozolomide repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection periodically for pharmacodynamic and pharmacokinetic correlative studies. Autophagic vesicles in blood samples are quantified by immunoblotting against the autophagy protein LC3 and by electron microscopy. Pharmacokinetics are analyzed by high-performance liquid chromatography with tandem mass spectrometry. Patients with tumors amenable to biopsy also undergo serial biopsies. Tumor tissue samples are assessed for tumor cell apoptosis and proliferation using Ki67 and TUNEL staining and for the number of autophagic vesicles and nuclear changes characteristic of apoptotic, autophagic, or necrotic cell death by western blotting and electron microscopy.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor

  * Metastatic or unresectable disease
  * Refractory to standard therapy or no standard therapy exists
* Measurable disease by RECIST criteria
* Brain metastases allowed provided patient completed radiotherapy (if radiotherapy was clinically indicated at the time of diagnosis) AND discontinued steroids prior to study enrollment

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,000/mm³
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 2.0 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN (< 3.0 times ULN in the presence of Gilbert's disease)
* AST and ALT ≤ 2.5 times ULN (≤ 5.0 times ULN in the presence of liver metastases)
* aPTT normal
* INR ≤ 1.5 (if on anticoagulation, INR must be < 1.5 prior to starting anticoagulation)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No porphyria
* No psoriasis, unless the disease is well controlled and patient is under the care of a specialist who agrees to monitor the patient for exacerbations
* No previously documented macular degeneration or diabetic retinopathy
* No concurrent serious illness including, but not limited to, any of the following:

  * Ongoing or active infection requiring parenteral antibiotics
  * Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, or unstable angina)
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Peripheral vascular disease ≥ grade 2 within the past year
  * Psychiatric illness/social situation that would limit compliance with study requirements
* No other concurrent malignancies, other than basal cell skin cancer, squamous cell skin cancer, carcinoma in situ of the cervix, or ductal or lobular carcinoma in situ of the breast

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* The following prior therapy is allowed in the adjuvant or metastatic disease setting:

  * Immunotherapy (interferon, aldesleukin, or sargramostim [GM-CSF])
  * Chemotherapy, either as a single-agent or as combination therapy
  * Vaccine therapy
  * Targeted or biological therapy
  * Chloroquine derivatives
* At least 4 weeks since prior active immunotherapy (aldesleukin, interferon, or ipilimumab)
* At least 4 weeks since prior chemotherapy
* At least 2 weeks since prior oral targeted therapies
* More than 4 weeks since prior and no other concurrent investigational anticancer therapy (except for vaccines)
* No prior temozolomide
* Prior radiotherapy allowed

  * If radiotherapy has been administered to a lesion, there must be radiographic evidence of progression of that lesion in order for that lesion to constitute measurable disease or to be included in the measured target lesions
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine, phenobarbital, primidone, or oxcarbazepine), rifampin, or Hypericum perforatum (St. John's wort)
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-06; Primary Completion 2011-07 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of hydroxychloroquine

SECONDARY OUTCOMES:
Toxicity rates
Pharmacodynamic and pharmacokinetic correlative endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Amaravadi, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States